CLINICAL TRIAL: NCT01699191
Title: Probiotics for the Treatment of Irritable Bowel Syndrome in Celiac Patients
Acronym: ProCel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Consultant in Gastroenterology, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ProCeDo
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: IBS in Celiac Desease
Keywords: Irritable Bowel Syndrome; Celiac Desease; Probiotic; Lactobacillus plantarum; Bifidobacterium breve; Lactobacillus casei; Bifidobacterium animalis
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic Mixture (Active Comparator): Probiotic mixture
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotic Mixture
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Probiotics play an important role in preventing overgrowth of potentially pathogenic bacteria and maintaining the integrity of the gut mucosal barrier. The beneficial effects of probiotics have been previously studied in adult patients with IBS. Clinical studies show that patients meeting the criteria for diagnosis for IBS have greater probability for being affected by celiac desease if compared to controls without IBS. Since one of the causes attributed to the onset of IBS is the modified flora gut, it is interesting to determine the beneficial effects that probiotics may have on gastrointestinal symptoms in celiac disease patients. The goal of the present study is to determine whether oral administration of a probiotic mixture of Lactobacillus plantarum 14D-CECT 4528, Lactobacillus casei, Bifidobacterium breve Bbr8 LMG P-17501, Bifidobacterium breve Bl10 LMG P-17500 and Bifidobacterium animalis under randomized, double-blind, placebo-controlled conditions would improve symptoms of adult celiac patients with IBS.

DETAILED DESCRIPTION:
This is a randomized, double blind study, placebo-controlled, carried out in three departments of gastroenterology in Southern Italy (Bari, Taranto e Castellana Grotte).

Celiac patients with Irritable Bowel Syndrome will considered eligible for inclusion. They will be between 18 and 65 years old and they will be in GFD for at least 2 year.

Will be excluded from the study patients with previous abdominal surgery, chronic disease, alarm signs of organic conditions, treatment with probiotics, prebiotics, antibiotics and antispasmodics in the previous month, immunodeficiency, pregnancy.

The size of the sample, which must show a benefit greater than 25% compared to placebo (untreated group that usually able to respond positive in 20% of cases), will require 58 patients per arm to ensure a power of 90% with an alpha error of 0.5.

Patient will be assigned consecutive numbers, starting with the lowest number available, and randomly assigned, with the use of a computer generated randomisation list using permuted block design, to receive orally either a probiotic mixture of Lactobacillus plantarum 14D-CECT 4528, Lactobacillus casei, Bifidobacterium breve Bbr8 LMG P-17501, Bifidobacterium breve Bl10 LMG P-17500 and Bifidobacterium animalis or placebo (sachets identical in taste and appearance to the active study product except for the absence of probiotic mixture) once a day.

The study consists of three phases:

1. phase of "running-in" of two weeks to reduce the possibility of a next significant placebo effect in which the patient should not take no product;
2. supplementation for 6 weeks in which the patient will take one packet per day of placebo or active product;
3. follow-up of 6 weeks.

Enrolled patients will be entered sequentially to receive the assigned treatment. Boxes containing placebo will have the same shape, dimension, indication and appearance as those containing the viable probiotic mixture and will be provided by the probiotic producer (Moviscom Srl, Rome, Italy) which ensure that the study is blinded for investigators and patients. Group assignment will be concealed from participants and investigators.

During the duration of the trial (w1- w14) patients will record gastrointestinal symptoms on weekly diary. During the same time will compiled, every two week, the Gastrointestinal symptom rating score (GSRS), that consists of a 15-point questionnaire to assess severity and frequency of symptoms validated by Svedlund et al.. For all patients will be collected, at T = 0 and T = 42 days, stool samples on which will be performed the extraction of DNA and RNA for a possible assessment of the intestinal microflora. Bacteria DNA in stools will be extracted and stored at -80°C for future analysis. At the end of the study, for patients who have achieved the primary objective will be made specific identification of the intestinal microflora for verify any amendments.

The compliance to the study will be demonstrated according to the number of sachets consumed by the patient during the 6 weeks of administration, and on the basis of the compilation of the questionnaires provided by the protocol.

Outcome Measures Primary outcome will be the incidence in IBS in celiac patients receiving probiotics as compared to those receiving placebo. We have chosen pain as the primary outcome measure, in line with the proposed points-to-consider for IBS trials.

IBS will be diagnosed and categorised according to ROME III criteria. Secondary outcomes are: 1) evaluation of frequency/severity of symptoms according to treatment arm; 2) modification of intestinal microbiota.

The analysis of the intestinal microbiota of these informative cases will help to assess whether there is a intestinal microbiota suggestive of future inset of IBS and ability of our probiotic mixture to stabilize the intestinal microbiota.

Adverse Events and Disallowed Medication Adverse events will be monitored throughout the study. Patients will not allowed to consume any probiotic other than those provided and they will be invited to continue their eating and physical exercise habits.

ELIGIBILITY:
Inclusion Criteria:

* Celiac patients aged between 18 and 65 years
* Diagnosis of IBS on the basis of Rome III criteria
* GFD
* Informed consent

Exclusion Criteria:

* Previous sigmoidoscopy or colonoscopy in the past 5 years
* Known concomitant organic diseases, including inflammatory bowel disease and other systemic diseases significant
* Treatment with antispasmodic drugs within the previous month
* Are pregnant
* Immunodeficiency
* Previous abdominal surgery, with the exception of the hernia repair or appendectomy
* Treatment with antibiotics within the previous month
* Treatment with probiotics and / or prebiotics within the previous month
* Participation in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Treatment of abdominal pain in celiac patients | 14 weeks
  Primary outcome will be the incidence in IBS in celiac patients receiving probiotics mixture as compared to those receiving placebo.
  IBS will be diagnosed and categorised according to ROME III criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ruggiero Francavilla, Principal Investigator — DEPARTMENT OF BIOMEDICINA ETA' EVOLUTIVA
Locations (1):
- Clinica Pediatrica, Bari, Apulia, Italy